CLINICAL TRIAL: NCT00754715
Title: A Phase I, Single-Centre, Randomised, Double-Blind, Placebo-Controlled Parallel-Group Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD2516 in Young and Elderly Healthy Volunteers After Oral Single Ascending Doses
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics After Single Doses of AZD2516 to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD, Medical Science Director, Emerging Analgesia, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D2080C00001; EudractCT: 2008-003598-42
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Healthy
Keywords: Multiple dosing study,; safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD2516 (Experimental)
  Interventions: Drug: AZD2516
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2516 — Solution administered once orally
  Arms: AZD2516
Drug: Placebo — Solution administered only once
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of AZD2516 following administration of a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy white males or non-fertile females between 20 to 45 years and 65 to 80 years old.
* Weight between 50 to 100 kg and a body mass index (BMI) between 19 to 28 kg/m2

Exclusion Criteria:

* History of previous or ongoing psychiatric disease.
* Abnormalities in ECG that may interfere with interpretation of data.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD2516 by assessment of serious adverse events, ECGs, vital signs and laboratory variables | From first to last visit

SECONDARY OUTCOMES:
Safety and tolerability of AZD2516 by assessment of non-serious adverse events | Collected from start of residential period until last visit.
Determine the single ascending dose pharmacokinetics of AZD2516 | PK sampling taken at defined timepoints during residential period

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fransson, MD, Principal Investigator — AstraZeneca; Lars Ståhle, MD, PhD, Study Chair — AstraZeneca
Locations (1):
- Research Site, Stockholm, Sweden